CLINICAL TRIAL: NCT05244694
Title: Impact of Insulin on Sympathetic Nervous System-mediated Peripheral Vasoconstriction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020286
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Vasoconstriction; Healthy; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insulin (Experimental): Participants will complete a 60 minute hyperinsulinemic-euglycemic infusion.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Priming dose then a constant infusion at 40 mU•m-2•min-1

SUMMARY:
The purpose of this project is to determine if hyperinsulinemia attenuates sympathetic nervous system-mediated vasoconstriction in the human leg.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult men and women;
* 18-45 years of age;
* BMI 18-30 kg/m2;
* non-pregnant/non-breastfeeding;
* non-nicotine users;

Exclusion Criteria:

* taking any medications known to affect metabolic, respiratory, cardiovascular, and/or autonomic functions

Self-reported history of:

* hepatic, renal, pulmonary, cardiovascular, or neurological disease;
* stroke or neurovascular disease;
* bleeding/clotting disorders;
* sleep apnea or other sleep disorders;
* diabetes;
* smoking;
* history of alcoholism or substance abuse, excessive alcohol consumption;
* hypertension;
* active cancer;
* autoimmune disease;
* immunosuppressant therapy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Amount of leg blood flow | Change from baseline at minute 60
  Measured with Doppler ultrasound (mL/min)

SECONDARY OUTCOMES:
Amount of muscle sympathetic nerve activity (MSNA) | Change from baseline at minute 60
  MSNA burst incidence (bursts/100 heart beats)
Amount of cerebral blood flow | Change from baseline at minute 60
  Measured with trans-cranial Doppler ultrasound (cm/s)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline L Limberg, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided